CLINICAL TRIAL: NCT05648825
Title: Transapical Beating-Heart Septal Myectomy for Symptomatic Nonobstructive Hypertrophic Cardiomyopathy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiang Wei (Other)
Responsible Party: Sponsor-Investigator, Xiang Wei, Division of Cardiothoracic and Vascular Surgery, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-S086
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Nonobstructive Hypertrophic Cardiomyopathy
Keywords: Septal Myectomy; Transapical Beating-heart Septal Myectomy; Minimally Invasive; Midventricular obstruction and cavity obliteration; Nonobstructive Hypertrophic Cardiomyopathy

STUDY DESIGN:
Intervention Model Description: Beating-Heart Myectomy Device
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transapical beating-heart septal myectomy (Experimental): Transapical beating-heart myectomy for the treatment of nonobstructive hypertrophic cardiomyopathy
  Interventions: Device: Transapical beating-heart septal myectomy

INTERVENTIONS:
Device: Transapical beating-heart septal myectomy — We have invented a beating-heart myectomy device. Using this device, myectomy could be performed in the beating heart via a mini-thoractomy approach. The whole process of resection is monitored, navigated, and evaluated by real-time transesophageal and transthoracic echocardiography. We are now conducting the study to explore the feasibility, the safety, and the efficacy of transapical beating-heart myectomy for the treatment of nonobstructive hypertrophic cardiomyopathy.

SUMMARY:
The primary purpose of this study is to evaluate the feasibility, the safety and the efficacy of the transapical beating-heart myectomy for the treatment of apical hypertrophic cardiomyopathy. This is a prospective, single-arm, single-center study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were diagnosed as nonobstructive hypertrophic cardiomyopathy, with maximal apical wall thickness ≥ 15 mm.
2. Patients with heart function of New York Heart Association ≥ class II.
3. Presenting with severe symptoms, e.g. angina, dyspnea, or fatigue, that were unresponsive or intolerant to pharmaceutical therapies;
4. Kansas City Cardiomyopathy Questionnaire (KCCQ) score < 80;
5. Presenting with one of the following conditions: midventricular obstruction with gradient ≥ 50 mmHg; grade II or higher diastolic dysfunction; apical aneurysm; ventricular tachycardia that needed an ICD implantation; pulmonary hypertension.
6. Patients who was informed the nature of the clinical trial, consented to participate in all of the activities of the clinical trial, and signed the informed consent form.

Exclusion Criteria:

1. Patients who were pregnant.
2. Patients who had concomitant diseases such as intrinsic valvular disease or coronary artery disease that needed open-chamber cardiac surgery.
3. Patients who had severe heart failure with left ventricle ejection fraction < 50%.
4. Patients whose estimated life expectancy < 12 months.
5. Patient who were non-compliant.
6. peak VO2 of cardiopulmonary exercise test ≥ 90% of predicted.
7. LVOT obstruction.
8. Patients under circumstances which were considered not suitable or prohibitive for participating the clinical trial at the discretion of the attending medical team and the researchers.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Procedural success | 6 months
  Kansas City Cardiomyopathy Questionnaire (KCCQ) score improvement of ≥10 points, New York Heart Association (NYHA) improvement ≥ 1 grade, stroke volume increased by ≥10 mL, and diastolic function grading at normal or grade I (of III) .

SECONDARY OUTCOMES:
Left ventricular end-diastolic pressure | 1 day
  Left ventricular end-diastolic pressure measure by hemodynamic catheterization.
Left ventricular end-systolic volume | 7 days and 6 months
  Left ventricular end-systolic volume and indexed by body surface area. A higher left ventricular end-systolic volume indicates enlarged left ventricular chamber.
Left ventricular end-diastolic volume | 7 days and 6 months
  Left ventricular end-diastolic volume and indexed by body surface area. A higher left ventricular end-diastolic volume indicates enlarged left ventricular chamber.
Obliteration | 6 months
  Rate of obliteration and ratio of obliteration to cavity as measured by TTE
Peak oxygen consumption | 6 months
  Peak oxygen consumption as measured by cardiopulmonary exercise testing.
pVO2 | 6 months
  pVO2 as measured by cardiopulmonary exercise testing.
Pulmonary artery wedge pressure | 3 days
  Pulmonary artery wedge pressure as measured by Swan-Ganz catheter.
Stroke volume | 3 days
  Stroke volume as measured by Swan-Ganz catheter.
Left ventricle mass | 6 months
  Left ventricle mass index (the ratio of left ventricle mass to body weight) as measured by cardiac magnetic resonance.
Cardiac diastolic function | 6 months
  The ratio between early mitral inflow velocity and mitral annular early diastolic velocity ( E/e') and ratio between early mitral inflow velocity and late mitral inflow velocity (E/A) as measured by transthoracic echocardiography.
Left atria volume | 6 months
  The left atria volume as measured by echocardiography.
Ventricular wall thickness | 6 months
  Ventricular wall thickness as measured by echocardiography.
LVOT gradient | 1 week, 6 months
  Resting and provoked left ventricular outflow tract gradient as measured by echocardiography.
Midventricular gradient | 1 week, 6 months
  Resting and provoked midventricular gradient as measured by echocardiography.
Device success | 6 months
  Successful accession, delivery, and retrieval of the resection device, successful resection of the ventricular myocardium, and free from conversion to midline thoracotomy during operation.
New York Heart Association class | 6 months
  New York Heart Association class, including grade I, grade II, grade III, grade IV. A higher grade means worse heart function.
6-minute walking test | 6 months
  6-minute walking test. A longer distance means better heart function.
Heart function-associated quality of life | 6 months
  Score of the Kansas City Cardiomyopathy Questionnaire. A higher score means better heart function.
Angina level | 6 months
  Score of the Seattle angina questionnaire.
NT-proBNP | N-terminal pro-brain natriuretic peptide
cTnI | 1 week, 6 months
  cardiac troponin I
Major adverse cardiovascular and cerebral events | 6 months
  Procedure-related mortality and unplanned surgical procedures during hospitalization, permanent pacemaker implantation, iatrogenic valvular injury, imaging examination-validated cerebral complications.
All cause mortality | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Wei, M.D., Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
All of the conclusive participant data, after removing the individual information of privacy, will be uploaded as supporting information when publishing the current study.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the current study is published.
Access Criteria: All readers who were interested in the current study.

REFERENCES:
- [Background] Fang J, Wang R, Liu H, Su Y, Chen J, Han X, Wei Y, Chen Y, Cheng L, Wei X. Transapical septal myectomy in the beating heart via a minimally invasive approach: a feasibility study in swine. Interact Cardiovasc Thorac Surg. 2020 Feb 1;30(2):303-311. doi: 10.1093/icvts/ivz249. PMID 31642911
- [Background] Schaff HV, Brown ML, Dearani JA, Abel MD, Ommen SR, Sorajja P, Tajik AJ, Nishimura RA. Apical myectomy: a new surgical technique for management of severely symptomatic patients with apical hypertrophic cardiomyopathy. J Thorac Cardiovasc Surg. 2010 Mar;139(3):634-40. doi: 10.1016/j.jtcvs.2009.07.079. PMID 20176208